CLINICAL TRIAL: NCT00573339
Title: Cardiac Magnetic Resonance Imaging Normal Reference Control Group Testing - Ancillary Study to Coronary Endothelial Function and Microvascular Disease in Women
Brief Title: Cardiac Magnetic Resonance Imaging (MRI) Normal Reference Control Group Testing
Status: Recruiting | Type: Observational
Sponsor: Cedars-Sinai Medical Center (Other)
Responsible Party: Principal Investigator, Noel Bairey Merz, Director, Cedars-Sinai Medical Center
Other Study IDs: IRB# 11753
Record Dates: First submitted 2007-12-13; First posted 2007-12-14 (Estimated); Last update posted 2023-09-01 (Actual); Status verified 2023-08

CONDITIONS: Healthy
Keywords: Cardiac; MRI; normal controls

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: None Retained — BUN and Creatinine blood tests
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Normal Controls
  Interventions: Other: Cardiac MRI

INTERVENTIONS:
Other: Cardiac MRI — up to 3 Cardiac MRI scans per participant in 1-4 months

SUMMARY:
The purpose of this research is to understand how to apply cardiac magnetic resonance imaging (CMR) to women with small artery heart disease by looking at the CMRs of women without heart disease. The investigators will study 40 women with no heart disease to learn more about the usefulness of CMR.

Women suffer more than men from this disorder of the small vessels compared to the large vessels. This results in delays in diagnosis, missed opportunities for treatment, and likely contributes to the increased death rate from heart disease in women compared to men. Current testing for small vessel disease is invasive and not performed routinely and women are often not initiated on appropriate lifesaving treatment. New imaging and noninvasive technology exists that may improve this situation. Imaging techniques such as cardiac magnetic resonance imaging (CMR) can now show the inner layers of the heart where the small vessel abnormality and myocardial ischemia exist. These techniques, while promising, have not been tested to determine if they can be used to diagnose and treat the small vessel coronary heart disease condition. They also have not been studied extensively in women without heart disease.

Gadolinium, the contrast agent that will be given Intravenously to all study participants during the cardiac MRI procedure, is contraindicated to patients with renal impairment. Even though it will only be given once to each of our patients, the investigators still wanted to establish the fact that these study participants have "normal" or good renal functioning by doing BUN and Creatinine blood tests prior to the administration of this contrast agent to their system. By adding these lab tests, the investigators will be more cautious to the well-being and safety of the study participants.

The investigators will be recruiting women aged 35-65 years with no known heart disease or heart disease risk factors like high blood pressure or high cholesterol. Participants will discuss the cardiac magnetic resonance procedure with a research doctor and if they agree, will fill out questionnaires related to their health, have blood draw and then undergo the CMR procedure. This can be completed in 1 or 2 visits. No follow up is needed.

DETAILED DESCRIPTION:
The women will be consented and enrolled. They will:

1. fill out baseline demographic and health history questionnaires;
2. have an exercise treadmill test (ETT) To rule out any underlying ischemic heart disease;
3. undergo rest-stress CMR testing (up to 3 scans);
4. peripheral arterial tonometry; and
5. have blood drawn for hematocrit, blood urea nitrogen (BUN),creatinine, and research protein quantitation with mass spectrometry and enzyme-linked immunosorbent assay (ELISA) for sensitive quantitation of cardiovascular biomarkers.
6. measure central arterial stiffness by noninvasive pulse wave analysis (PWA) using SphygmoCor (done up to 3 times-once at each MRI visit).

ELIGIBILITY:
Inclusion Criteria:

1. Women without signs and symptoms of myocardial ischemia (chest pain, abnormal stress testing, abnormal noninvasive testing).
2. No cardiac risk factors by Framingham/NCEP criteria, age and BMI matched to the Cardiac Syndrome X population, and a normal exercise stress test.

Exclusion Criteria:

1. Contraindications to CMR testing (metal devices in chest, claustrophobia, known angioedema).
2. Contraindication to Adenosine or Lexiscan (regadenoson) including heart block (second and third degree) and sinus node disease, significant COPD/asthma, or systemic hypotension (<90 mmHg).
3. Contraindication to Dobutamine including severe systemic hypertension (≥ 220/120 mmHg), unstable angina, significant aortic valve stenosis, complex cardiac arrhythmia including uncontrolled atrial fibrillation, hypertrophic obstructive cardiomyopathy, myocarditis, endocarditis, pericarditis, or uncontrolled congestive heart failure.
4. Contraindication to Gadolinium (renal impairment).
5. Any renal disease.
6. Pregnant and lactating women.
7. Inability to perform exercise, eg. orthopedic limitations.
8. Allergy to animal dander.

Ages: 35 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Healthy women
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2007-05; Primary Completion 2030-12 (Estimated); Study Completion 2030-12 (Estimated)

PRIMARY OUTCOMES:
Cardiac MRI | at study visit

CONTACTS AND LOCATIONS:
Overall Officials: C. Noel Bairey Merz, MD, Principal Investigator — Cedars-Sinai Medical Center
Locations (1):
- Cedars-Sinai Women's Heart Center, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: Yes